CLINICAL TRIAL: NCT00334113
Title: Telerehabilitation Intervention to Promote Exercise for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F4202-I
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Diabetes Mellitus; Exercise; Obesity; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Participants in this arm will meet with an exercise physiologist and obtain an exercise prescription for a walking program. In addition, they will recieve an intervention that will be delivered over an automated telephone system (TLC-PED). These automated phone calls with voice response and voice recognition capabilities will occur weekly over a 6 month period. During these calls, participants' physical activity will be monitored, new physical activities goals will be set, information about physical activity and the associated health benefits will be provided, and barriers to physical activity will be explored.
  Interventions: Behavioral: TLC-PED
- Arm 2 (No Intervention): This is the "treatment as usual" condition. Participants in this condition will also have 2 sessions with an exercise physiologist and will receive an exercise prescription for a home based walking program. The will not receive the automated phone calls each week that are designed to motivate physical activity.

INTERVENTIONS:
Behavioral: TLC-PED — Telephone-Linked Care - Promoting Exercise for Diabetes (TLC-PED), a method that uses interactive voice response and speech recognition technologies, will be developed to provide individualized and personalized motivational messages using automated telephone calls for veterans with Type 2 diabetes who participate in a home based walking program.
  Arms: Arm 1

SUMMARY:
The overarching objective of this study is to develop an innovative strategy to address the problems of obesity and diabetes by promoting exercise adoption. An automated telephone intervention will be developed that can be used to enhance exercise adoption over a twelve month period in a population of overweight or obese veterans with Type 2 diabetes.

DETAILED DESCRIPTION:
Approximately two thirds of American adults are overweight (body mass index - BMI > 25), and nearly one third of American adults are obese (BMI > 30) with veterans exhibiting even higher rates of being overweight and obese than those in the general population. Obesity is a significant risk factor for a number of serious medical conditions, including diabetes, and is associated with high rates of morbidity, and mortality. Greater than 80% of individuals with diabetes are overweight or obese. Sixteen million Americans have been diagnosed with diabetes, and it has been speculated that this number will increase to 23 million by the year 2010. Furthermore, there is a substantially higher prevalence of diabetes in the veteran population as compared to the general population, with nearly 16 percent of veterans being affected. This alarming increase has been associated with the increasing prevalence of obesity and sedentary lifestyles. In a conference conducted by the National Institute of Diabetes and Digestive and Kidney Diseases in 1999, it was concluded that a major research initiative was needed to address the growing problem with physical inactivity and obesity because of the major impact these behaviors have on the development and treatment of diabetes.

The benefits associated with exercise in the diabetic population are extensive, and even though regular exercise is typically prescribed as a significant component of the diabetic treatment plan, compliance tends to be very poor. The overarching objective of this study is to adapt a low cost telephone intervention to be used to enhance exercise adoption in a population of overweight or obese veterans with type 2 diabetes. The primary aim of this study is to implement and evaluate the effectiveness of this telehealth intervention over a six month period. The secondary aim is to evaluate the impact this telehealth intervention has on weight and other diabetes relevant physical health parameters, quality of life and psychological distress. If the telehealth intervention is found to be efficacious, the tertiary aim will be to evaluate the cost effectiveness of the intervention. Over a 4-year period, 140 overweight or obese veterans with type 2 diabetes will be recruited from the VA Boston Healthcare System. All participants will be evaluated and provided with an exercise prescription for a home based walking program. Participants will be randomized to either the Exercise Prescription condition alone, or Exercise Prescription plus TLC-PED (Telephone Linked Care - Promoting Exercise for Diabetes), an automated telehealth intervention. TLC-PED will use interactive voice response and recognition telephone technology to provide individualized phone messages for participants with diabetes. It will be developed to incorporate theoretical principles that are known to enhance exercise adoption. Specifically, the intervention will use motivating principles based on the transtheoretical model of change. Those in the TLC-PED condition will receive weekly automated telephone calls for a six month period. It is hypothesized that overweight veterans with diabetes who receive the TLC-PED intervention (versus those who do not) during their six month participation in a home based walking program will be more likely to engage in regular physical activity and obtain improvements in self-reported physical activity, and maintain these changes over a twelve month period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus
* Receive a medical clearance from physician
* Be sedentary
* Be interested in exercising
* Have a BMI > 25 kg/m2
* Have an HbA1c between 7 & 10%
* Be on medication for diabetes

Exclusion Criteria:

* Significant peripheral neuropathy
* Active psychosis
* Psych admission or substance abuse in the last 6 months
* Severe brain dysfunction
* Abnormal ECG
* Orthopedic related limitations
* Unable to understand English
* No direct access to telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Mori, PhD, Principal Investigator — VA Medical Center, Jamaica Plain Campus
Locations (1):
- VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts, United States

REFERENCES:
- [Result] Seligowski AV, Pless Kaiser AP, Niles BL, Mori DL, King LA, King DW. Sleep quality as a potential mediator between psychological distress and diabetes quality of life in veterans with type 2 diabetes. J Clin Psychol. 2013 Oct;69(10):1121-31. doi: 10.1002/jclp.21866. Epub 2012 May 25. PMID 22638910

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 89 participants were enrolled in this study, only 66 participants were randomized. Of the difference, 18 were determined to be ineligible (17 for medical reasons, 1 for other reasons), and 5 participants dropped out before randomization.
Groups:
- TLC-PED: Participants in this arm will meet with an exercise physiologist and obtain an exercise prescription for a walking program. In addition, they will be called every week by an automated telephone system that is designed to motivate individuals with type 2 diabetes to participate in regular physical activity.
  Motivate physical activity in diabetic individuals.: Telephone-Linked Care - Promoting Exercise for Diabetes (TLC-PED), a method that uses interactive voice response and speech recognition technologies, will be developed to provide individualized and personalized motivational messages using automated telephone calls for veterans with Type 2 diabetes who participate in a home based walking program.
- Treatment as Usual: This is the "treatment as usual" condition. Participants in this condition will also have 2 sessions with an exercise physiologist and will receive an exercise prescription for a home based walking program. The will not receive the automated phone calls each week that are designed to motivate physical activity.
Period: Overall Study
Arm/Group | TLC-PED | Treatment as Usual
Started | 32 | 34
Completed | 30 | 31
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TLC-PED | Treatment as Usual | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 62 (11) | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 1 | 2 | 3
7 Day Physical Activity Recall [Mean (Standard Deviation); unit: minutes of physical activity in a week] | 370 (251) | 341 (329) | 355 (339)

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Physical Activity Recall (PAR)
Description: A self-report measure of minutes of physical activity over the previous 7 days.
Time Frame: six months
Population: Participants analyzed varies from completed participants since the completed number comes from those who stayed in the study through the 12 months (6 months post intervention). In TAU, the number who completed exceeds the number analyzed since 1 participant did not show for the 6 month assessment but did show for the 12 month follow up assessment.
Measure: Mean (Standard Deviation); unit: minutes per week
Groups:
- TLC-PED: Participants in this arm will meet with an exercise physiologist and obtain an exercise prescription for a walking program. In addition, they will be called every week by an automated telephone system that is designed to motivate individuals with type 2 diabetes to participate in regular physical activity.
Arm/Group | TLC-PED | Treatment as Usual
Number analyzed (Participants) | 32 | 30
minutes per week | 319 (251) | 360 (329)

ADVERSE EVENTS:
Arm/Group | TLC-PED | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 5/32 | 6/34
Other Adverse Events (participants affected / at risk) | 8/32 | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TLC-PED (N=32) | Treatment as Usual (N=34)
Cardiac symptoms (Cardiac disorders) | 1 | 4 — Various symptoms including angina, chest pain, MI
UTI (Renal and urinary disorders) | 1 | 0 — UTI that resulted in hospitalization
hypoglycemia that resulted in hospitalization (Endocrine disorders) | 3 | 0
fever of unknown origin that resulted in hospitalizaton (Infections and infestations) | 1 | 0
tonsillar cancer that resulted in hospitalizaton (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
small stroke that resulted in hospitalization (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TLC-PED (N=32) | Treatment as Usual (N=34)
orthopedic pain/injury (Musculoskeletal and connective tissue disorders) | 6 | 2 — various pains in legs and feet were reported
bronchitis/pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes